CLINICAL TRIAL: NCT06607276
Title: A Phase 2, Randomized, Controlled, Multicenter Study of Adjuvant Adebrelimab Combined With Capecitabine in Resected Cholangiocarcinoma With High-risk Factors: ACHIEVE
Brief Title: Phase 2 Trial of Adjuvant Adebrelimab Combined With Capecitabine in High-Risk Resected Cholangiocarcinoma: ACHIEVE
Acronym: ACHIEVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jinling Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-571
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cholangiocarcinoma Cancer; Adebrelimab (SHR-1316)
Keywords: Adebrelimab; capecitabine; Cholangiocarcinoma; Adjuvant Therapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adebrelimab and capecitabine (Experimental)
  Interventions: Drug: Adebrelimab and capecitabine
- capecitabine (Active Comparator)
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: Adebrelimab and capecitabine — Adebrelimab: 1200mg, IV, q3w for one year; capecitabine:1250mg/m2, po, bid,d1-14, q3w, for 6-8 cycles
  Arms: Adebrelimab and capecitabine
Drug: capecitabine — capecitabine:1250mg/m2, po, bid,d1-14, q3w, for 6-8 cycles
  Arms: capecitabine

SUMMARY:
Biliary tract malignancies (BTC) are malignant tumors that originate from the epithelium of the bile ducts. Currently, the optimal treatment for biliary tract malignancies is radical surgical resection. In recent years, with the advancement of imaging technology and surgical techniques, there has been certain progress in the diagnosis and treatment of biliary tract malignancies. However, the surgical resection rate and long-term survival rate after surgery are still not satisfactory, and the high postoperative recurrence rate is an important factor affecting the long-term survival of patients. Therefore, there is an urgent need to explore new postoperative adjuvant treatment plans to reduce postoperative tumor recurrence, which is of great significance for extending the survival of patients with biliary tract malignancies. In the NCCN and CSCO guidelines, capecitabine is listed as a category I recommendation for adjuvant treatment of biliary tract malignancies (BTC). However, in clinical practice, the use of capecitabine or tegafur for postoperative patients with cholangiocarcinoma at high risk of recurrence still has a high recurrence rate. Therefore, there is still a huge unmet need in the clinical adjuvant treatment after surgery for biliary tract malignancies. Based on the above background, we plan to carry out a randomized, open, and comparative study to observe the efficacy and safety of Adebrelimab combined with capecitabine for adjuvant treatment in patients with biliary tract malignancies after surgery, and to explore treatment methods to improve the efficacy of postoperative adjuvant treatment for cholangiocarcinoma.

DETAILED DESCRIPTION:
Postoperative adjuvant therapy for biliary system tumors has long lacked a universally recognized standard regimen. The BILCAP trial results showed a survival benefit with adjuvant therapy. The BILCAP study filled the gap in the field of postoperative adjuvant therapy for biliary system tumors. In the study, the median overall survival (OS) in the capecitabine group was 51.1 months, compared to 36.4 months in the observation group. The median recurrence-free survival (RFS) in the capecitabine group was 24.4 months, compared to 17.5 months in the observation group. Compared to the observation group, adjuvant therapy with capecitabine significantly prolonged both OS and RFS, and the capecitabine group had good tolerability with no chemotherapy-related deaths. In addition, the ASCOT study reported that adjuvant therapy with tegafur after surgery could prolong the RFS rate in patients. Therefore, in the NCCN and CSCO guidelines, capecitabine is listed as a category I recommendation for adjuvant therapy of biliary tract malignancies (BTC). However, it is regrettable that the latest reports show that in the intention-to-treat (ITT) population, the BILCAP trial failed to reach its primary endpoint of OS, with the median OS in the study group and the control group being 51.1 months and 36.4 months, respectively [HR=0.81, 95% CI(0.63,1.04), P=0.097]. Furthermore, in clinical practice, the use of capecitabine or tegafur after surgery in patients with cholangiocarcinoma at high risk of recurrence still has a high recurrence rate. Therefore, there is still a significant unmet need in the clinical postoperative adjuvant therapy for biliary tract malignancies.Based on the above background, we plan to carry out a randomized, open, and comparative study to observe the efficacy and safety of Adebrelimab combined with capecitabine for adjuvant treatment in patients with biliary tract malignancies after surgery, and to explore treatment methods to improve the efficacy of postoperative adjuvant treatment for cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign an informed consent form;
2. Ages 18-75, both genders eligible;
3. ECOG performance status score (PS score) of 0 or 1;
4. Patients with histologically confirmed cholangiocarcinoma (including intrahepatic cholangiocarcinoma and hilar cholangiocarcinoma), who have undergone R0 resection and have high-risk factors for recurrence;

   High-risk factors are defined as follows:

   Intrahepatic cholangiocarcinoma ( Single tumor > 5 cm, multiple tumors, liver capsule breach, vascular invasion, regional lymph node metastasis) Hilar cholangiocarcinoma (Tumor invasion into surrounding tissues, vascular invasion, regional lymph node metastasis)
5. No evidence of recurrence or metastatic lesions on imaging within 28 days prior to randomization;
6. No prior systemic anti-cancer therapy (including radiotherapy, chemotherapy, targeted therapy, immunotherapy) before curative resection;
7. Laboratory test values within 7 days prior to the first dose of study medication meet the following criteria:

   Complete blood count: (except for hemoglobin, no blood transfusion or use of granulocyte colony-stimulating factor [G-CSF], no medication correction within 2 weeks prior to screening):

   Absolute neutrophil count ≥1.5×109/L; Platelets ≥75×109/L; Hemoglobin ≥90 g/L;

   Biochemical tests:

   Serum albumin ≥30g/L; Serum total bilirubin ≤1.5×ULN; ALT and AST ≤3×ULN; Serum creatinine ≤1.5×ULN; or Cr clearance rate >50 mL/min International normalized ratio (INR) ≤1.2 or prothrombin time (PT) exceeding the normal control range by ≤2 seconds; Urine protein <2+ (if urine protein ≥2+, a 24-hour (h) urine protein quantification can be performed, and a 24h urine protein quantification of <1.0g is eligible for enrollment);
8. Life expectancy of more than 6 months.

Exclusion Criteria:

1. Pathological diagnosis of mixed hepatocellular carcinoma and other non-hepatic extra-bile duct cholangiocarcinoma or ampulla of Vater malignant tumor components;
2. History of prior systemic treatment;
3. History of or concurrent other malignancies, excluding non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid carcinoma that have been adequately treated;
4. Active tuberculosis infection. Patients with active tuberculosis infection within 1 year prior to enrollment; history of active tuberculosis infection more than 1 year prior to enrollment without proper anti-tuberculosis treatment or tuberculosis is still active;
5. History of autoimmune diseases or immunodeficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, or multiple sclerosis;
6. Requirement for long-term systemic corticosteroids (dosage equivalent to >10mg prednisone/day) or any other form of immunosuppressive treatment. Subjects using inhaled or topical corticosteroids may be included;
7. Severe cardiopulmonary or renal dysfunction;
8. Inadequately controlled arterial hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) (based on the average of ≥2 blood pressure readings), allowing the achievement of the above parameters through the use of antihypertensive treatment; history of hypertensive crisis or hypertensive encephalopathy;
9. Within 3 months prior to enrollment, significant clinical bleeding symptoms or a clear tendency to bleed; abnormal coagulation function (PT >14s), tendency to bleed, or undergoing thrombolytic or anticoagulant therapy;
10. HBV DNA >2000 IU/ml, active HCV infection (positive HCV antibody and HCV-RNA level above the lower limit of detection);
11. Active infection requiring systemic treatment;
12. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive;
13. History of psychiatric medication abuse, alcoholism, or drug addiction;
14. History of allergy to study medication;
15. Other factors deemed by the investigator to potentially affect subject safety or trial compliance. Such as severe diseases requiring concurrent treatment (including psychiatric diseases), severe laboratory test abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
one year recurrence free survival rate (1-year RFS) | 1 year
  1-year RFS refers to the proportion of patients who have not experienced disease recurrence or death within one year from randomization.

SECONDARY OUTCOMES:
overall survival (OS) | 3 year
  Overall survival (OS) refers to the length of time from randomization until death from any cause.
Recurrence free survival (RFS) | 2 year
  Recurrence-free survival (RFS) refers to the length of time after randomization during which a patient remains free from the recurrence of the disease.
minimal residual disease (MRD) | 2 year
  MRD refers to tumor-derived molecular abnormalities that are undetectable by imaging or traditional laboratory methods after treatment, but can be identified through liquid biopsy.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Jinling Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yancheng NO.1 People's Hospital, Yancheng, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Cheng Y, Zhang Y, Li C, Li X. Adebrelimab plus capecitabine versus capecitabine monotherapy for adjuvant treatment of high-risk resected cholangiocarcinoma (ACHIEVE): protocol for a phase II, multicentre, randomised controlled trial. BMJ Open Gastroenterol. 2025 Jul 30;12(1):e001892. doi: 10.1136/bmjgast-2025-001892. PMID 40738506